CLINICAL TRIAL: NCT00720720
Title: Effect of Phytosterols Enriched Products Consumption on Carotid Artery Artherosclerotic Plaque
Acronym: PHYTOPLAQUES
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment and organizational difficulties
Sponsor: French Cardiology Society (Other)
Collaborators: Fondation Coeur et Artères (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2006-03
Record Dates: First submitted 2008-07-21; First posted 2008-07-23 (Estimated); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): plant sterol enriched margarine
  Interventions: Dietary Supplement: plant sterol enriched margarine
- 2 (Placebo Comparator): placebo margarine
  Interventions: Dietary Supplement: plant sterol enriched margarine; Dietary Supplement: placebo margarine

INTERVENTIONS:
Dietary Supplement: plant sterol enriched margarine — Each group will have to consume 20 grams of margarines (either placebo or enriched in plant sterols) in one or two catches per day, for 8 weeks.
Dietary Supplement: placebo margarine
  Arms: 2

SUMMARY:
The objective of this exploratory study is to analyse in humans any qualitative changes of carotid artery atherosclerotic plaque under the influence of plant sterols consumption.

ELIGIBILITY:
Inclusion Criteria:

* Patient, men and women, aged between 40 to 75 ans (limits included) willing to participate to the study and have signed informed consent for its participation in the study
* Displaying a non serious chirurgical indication of clinical asymptomatic carotid stenosis defined by:

  * atherosclerotic stenosis of 60 to 75% on one on the two carotid junction (external carotid excluded) according to criteria from NASCET
  * without constituted or transitory recent cerebral vascular accident. The discovery of an ischaemic after-effect on a systematic scanner is not a criterion of exclusion
* Subject with normal body weight or in over weight (Body Mass Index ranged between 19 and 30 kg/m2, [limits included])
* Subject willing to follow dietary recommendations advised during hypercholesterolemia (according to AFSSAPS' recommendations)
* Subject with social insurance or equivalent.

Exclusion Criteria:

* Subject who, according to AFSSAPS' recommendations, should received a hypocholesterolemic therapy before the end of the study.
* Subject with a history of diabetes
* Subject with cardiac disease such as unstable angina, myocardial infarction, coronary angioplasty, coronary artery bypass graft surgery, or moderate or severe congestive heart failure within the last 6 months.
* Subject with plasma triglyceride levels higher than 2,5 g/l [limit included],
* Subject taking any drugs known to affect the evaluation of studied parameters
* Subject with severe or acute disease that could affect the results of the study or subject safety
* Subject with regular consumption of phytosterol enriched foods products during the study.
* Subject with any other medical condition or laboratory abnormality prior to recruitment that in the opinion of the principal investigator could affect subject safety or render unlikely trial to be conducted to the end.
* For women: pregnancy or breast feeding or subject likely to be pregnant during the study.
* For women: subject likely to modify their hormonal therapy during the study
* Subject in exclusion period after its participation in an other clinical trial

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-12-16 (Actual); Primary Completion 2010-02-24 (Actual); Study Completion 2010-02-24 (Actual)

PRIMARY OUTCOMES:
Effect of Phytosterols Enriched Products Consumption on Carotid Artery Artherosclerotic Plaque | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eric BRUCKERT, PU PH, Principal Investigator — APHP
Locations (3):
- France (3):
  - Hôpital cardio-vasculaire et pneumologique Louis Pradel, Bron
  - Clinique d'Endocrinologie, Maladies Métaboliques et Nutrition, Nantes
  - Groupe Hospitalier Pitié-Salpêtrière, Endocrinology and Metabolism Department, Paris